CLINICAL TRIAL: NCT00436605
Title: A Phase 2 Study of Dasatinib in Advanced Melanoma
Brief Title: Dasatinib in Treating Patients With Stage III Melanoma That Cannot Be Removed By Surgery or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00219; NCI-2009-00219 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000528937; UMN-2007UC009; YALE-HIC-0608001765; HIC#0608001765 (Other: Yale University); 7758 (Other: CTEP); P30CA016359 (NIH)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2011-10

CONDITIONS: Recurrent Melanoma; Stage IIIA Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Dasatinib

ARMS (1):
- Treatment (kinase inhibitor therapy) (Experimental): Patients receive oral dasatinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib
  Other Names: BMS-354825; Sprycel

SUMMARY:
This phase II trial is studying how well dasatinib works in treating patients with stage III melanoma that cannot be removed by surgery or stage IV melanoma. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with stage III unresectable or stage IV melanoma treated with dasatinib.

II. Determine the progression-free survival of patients treated with this drug.

SECONDARY OBJECTIVES:

I. To assess the expression of targets of Dasatinib prior to treatment by obtaining pre-treatment biopsies or examining paraffin-embedded tissues from previous tumor resections.

II. In selected patients (approximately 5-10) where tumor tissue is available pre-treatment and can be obtained post-treatment with Dasatinib (21 days after initiation of therapy), to determine if Dasatinib induces changes in expression of selected targets and downstream mediators, including MEK, ERK and RSK-1.

III. To assess toxicity.

OUTLINE:

Patients receive oral dasatinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage III unresectable or stage IV melanoma
* Measurable disease
* Must have evidence of tumor growth or new lesions within the past 6 months
* No large pleural effusions
* No known brain metastases or leptomeningeal metastases

  * Previously treated brain metastases allowed provided there is no requirement for steroids AND no evidence of progression for ≥ 8 weeks after treatment
* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Life expectancy > 3 months
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL (transfusions allowed)
* Bilirubin ≤ 1.5 mg/mL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* PT/INR and PTT normal
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* No medical condition that may affect the ability to swallow and retain dasatinib tablets, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication
  * Requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* No clinically significant cardiovascular disease, including any of the following:

  * Myocardial infarction or ventricular tachyarrhythmia within the past 6 months
  * Prolonged QTc > 480 msec
  * Major conduction abnormality (unless a cardiac pacemaker is present)
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * History of significant congenital or acquired bleeding disorder, including any of the following:

    * Von Willebrand's disease
    * Antifactor VIII antibodies
  * Dyspnea at rest or with minimal exertion
  * Uncontrolled seizure disorder
  * Psychiatric illness or social situations that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other active malignancy within the past 3 years except curatively treated stage I malignancies or resected skin carcinomas
* Recovered from prior therapy
* Prior adjuvant therapy for stage II or III melanoma allowed
* No prior cytotoxic therapy for metastatic melanoma
* No prior dasatinib or other inhibitors of src, bcr-abl, c-Kit, EPHA2, and PDGFRβ
* No more than 2 prior immunomodulator therapies for metastatic melanoma
* At least 1 week since prior and no concurrent warfarin or other anticoagulants or medications that inhibit platelet function (including acetylsalicylic acid)
* At least 1 week since prior and no concurrent steroids or other immunosuppressive agents

  * Concurrent steroids to treat induced pleural effusions allowed
* At least 3 weeks since prior immunomodulators including, but not limited to, any of the following:

  * Aldesleukin
  * Cancer vaccines
  * T-cell-activating monoclonal antibodies
* At least 4 weeks since prior radiotherapy

  * Prior palliative radiotherapy to a single site of disease allowed (tumor is not considered evaluable for response unless there is tumor progression at the site of radiation)
* More than 7 days since prior and no concurrent CYP3A4 inhibitors
* At least 7 days since prior and no concurrent agents with proarrhythmic potential
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies
* No concurrent enzyme-inducing anticonvulsant agents
* No concurrent grapefruit or grapefruit juice
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent CYP3A4 inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-12; Primary Completion 2010-03 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Kluger, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Started | 39
Completed | 36
Not Completed | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Full Range); unit: years] | 64 [37 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Objective Response(Partial Response and Complete Response) as Measured by RECIST Criteria
Description: Only those patients who have measurable disease present at baseline, have received at least one course of therapy, and have had their disease re-evaluated will be considered evaluable for response. A Simon's optimum two-stage design will be used.
Time Frame: After every 8 weeks (or 2 courses), assessed up to 4 weeks after completion of treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 36
participants | 2

2. Primary Outcome: Progression-free Survival
Description: Progression will be evaluated in this study using the new international criteria proposed by the RECIST Committee. A Simon's optimum two-stage design will be used
Time Frame: Time from start treatment to time of progression, assessed up to 6 months
Measure: Mean (Full Range); unit: weeks
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 36
weeks | 8 [3 to 136]

ADVERSE EVENTS:
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 20/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Kinase Inhibitor Therapy) (N=39)
Fatigue (General disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Anorexia (General disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Kinase Inhibitor Therapy) (N=39)
Fatigue (General disorders) | 30
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 27
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 14
Nausea (Gastrointestinal disorders) | 26
Emesis (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 14
Weight Loss (General disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 17
Pruritis (Skin and subcutaneous tissue disorders) | 7
Anorexia (General disorders) | 23
Xerostomia (General disorders) | 13
Heartburn (Gastrointestinal disorders) | 6
Taste Alternation (Gastrointestinal disorders) | 8
Edema (Vascular disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less